CLINICAL TRIAL: NCT07369180
Title: Safety and Efficacy of an Accelerated, Rectangular Waveform rTMS Protocol in Treatment of Adults With Major Depressive Disorder.
Brief Title: NQ Square TMS for MDD 1Dx3S Adults Multi-site Sham-controlled Protocol
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroQore Inc. (Industry)
Collaborators: Makromed Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-NQ-2025-01; BRANY IRB File #2-02-5-1959 (Other: Biomedical Research Alliance of New York (BRANY))
Record Dates: First submitted 2026-01-24; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
Keywords: Maor Depressive Disorder (MDD); Accelerated Treatment; 1-day Treatment
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly and in double-blind manner (blind to investigator and participant) provided the active or sham treatment with NeuroQore's TMS system using a neuro-navigation system utilizing MRI to identify individualized target area for stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Device operators delivering the treatment regimen are also masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Accelerated Protocol (Experimental): Three 19-min TMS treatment protocol delivered on the same day, with 1 hour rest between the sessions.
  Interventions: Device: Active Accelerated rTMS Treatment
- Sham Accelerated Protocol (Sham Comparator): Three 19-min TMS treatment protocol simulated but blocked from delivery to the target region in Cortex, on the same day, with 1 hour rest between the sessions.
  Interventions: Device: Sham Accelerated rTMS Treatment

INTERVENTIONS:
Device: Active Accelerated rTMS Treatment — 1 Day x 3 Sessions of 19-minutes active rTMS treatment, with 60 minutes rest between sessions.
  Arms: Active Accelerated Protocol
Device: Sham Accelerated rTMS Treatment — 1 Day x 3 Sessions of 19-minutes sham rTMS treatment, with 60 minutes rest between sessions. It simulates the treatment regimen but blocks the treatment from reaching the target in Cortex.
  Arms: Sham Accelerated Protocol

SUMMARY:
Transcranial Magnetic Stimulation (TMS) Therapy is a non-invasive procedure that uses magnetic pulses to stimulate the cortex (brain) to treat Major Depressive Disorder (MDD). Currently established therapy uses one 19-minute treatment session per day for 5 days per week for 6 weeks, for a total of 30 treatment sessions.

The goal of this multi-site sham-controlled double-blinded randomized clinical trial is to evaluate the safety and effectiveness of accelerating the delivery of the NeuroQore Square TMS system's rectangular waveform rTMS protocol for the treatment of adults aged 22-85 with Major Depressive Disorder.

The accelerated protocol of this study will involve the same currently FDA-cleared 19-min treatment session offered three times in a single day, with no additional treatment sessions.

DETAILED DESCRIPTION:
Study Description:

This multi-site sham-controlled double-blinded randomized study will evaluate the safety and efficacy of accelerating the delivery of the NeuroQore Square TMS system's rectangular waveform rTMS protocol for the treatment of adults aged 22-85 with Major Depressive Disorder.

Currently cleared protocol with the FDA (the Standard of Care Protocol) is one 19-min treatment session a day for 5 days/week for 6 weeks. The accelerated protocol will involve the same 19-min treatment session offered three times in a single day, with no additional treatment sessions.

Primary Objectives:

1. To assess the efficacy of the NeuroQore Square TMS system, with accelerated delivery, in the treatment of adults with major depressive disorder as measured by a change in MADRS score 24 hours, 7 days and 30 days after the treatment end.
2. To compare the safety profile of the accelerated delivery protocol to the historical safety profile of the Standard of Care protocol.

End Points:

Primary

* Change in MADRS score from baseline to 24 hours, 7 days and 24 days post treatment.
* Number and type of adverse events.

Secondary

* Change in PHQ-9 score from baseline to 24 hours, 7 days and 24 days post treatment.

Study Population:

Men and women 22-85 with major depressive disorder that have failed one medication in the current episode. Its demographics will reflect variations in race, ethnicity, residence status (urban, suburban, rural), and socioeconomic status (education, profession).

Study Intervention:

NeuroQore TMS System includes (1) a pulse generator, (2) a magnetic coil, (3) a coil cooler, and (4) a chair with a headpiece. It has been cleared for clinical use (K232688) by the FDA for the treatment of Major Depressive Disorder (MDD) using a 19-min Standard of Care protocol.

Treatment during this study will be administered according to this protocol and following the instructions in the device user manual. Personalized stimulation targets will be produced from participants' structural MRI via the proprietary targeting generation component of the NeuroQore TMS system.

Only personnel trained and certified by NeuroQore will be permitted to administer treatment. All session and device information will be captured on appropriate data collection forms.

Study Duration:

The study is anticipated to last up to 3 months including enrollment and follow-up.

Individual participant duration in the study will be 1 day of treatment, 24- hour, 7-day and 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 22-85.
2. Current diagnosis of major depressive disorder according to the criteria defined in the current Diagnosis and Statistical Manual of Mental Disorders (DSM-V) without psychotic features. The diagnosis of DSM-5 criteria-defined MDD will be made by a psychiatrist in light of a comprehensive psychiatric evaluation and other available clinical data.
3. Drug-resistant MDD (lack of improvement on antidepressant medication in the current episode, despite adequate dose and duration and adherence to treatment).
4. MADRS score > 20 at baseline and immediately prior to the day of treatment.
5. Agrees to adhere to the study treatment and follow-up schedule.
6. Evidence of no change in AD medications or psychotherapy from 4 weeks prior to enrollment and participant's agreement not to request such changes through 2 weeks after study regimen treatment.
7. Fluent in English.

Exclusion Criteria:

1. Any medical conditions that would preclude the use of rTMS to treat depression.
2. Any conditions that would prevent the ability to undergo MRI testing.
3. Pregnancy as determined by serum/urine pregnancy test
4. History of epilepsy, seizure(s), or a seizure disorder as determined by the principal investigator based on a medical history obtained from the patient and/or others authorized to provide such history, combined with a brief screening instrument.
5. Active substance abuse
6. Diagnosis of bipolar or psychotic disorder
7. Considered to be at moderate-high risk of suicide according to the C-SSRS assessment (i.e., Answers YES to Question 3 and NO to Question 6; or answers YES to Question 4, 5, or 6)
8. As determined by the Principal Investigator, subjects with cognitive impairment according to either the medical history obtained from the patient and/or a reliable secondary source, or the results of the Montreal Cognitive Assessment (MoCA) performed during screening.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
MADRS Score | From enrollment to final MADRS score assessment within 6 weeks.
  Change in MADRS score from baseline to immediately post treatment, 24 hours, 7 days and 30 days post-treatment.

SECONDARY OUTCOMES:
PHQ-9 Score | From enrollment to final PHQ-9 score assessment within 6 weeks.
  Change in PHQ-9 score from baseline to immediately post treatment, 24 hours, 7 days and 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ramgopal, DO, Principal Investigator — LGTC Group
Locations (2):
- United States (2):
  - LGTC Group, Campbell, California
  - LGTC Group, Sunnyvale, California

IPD SHARING:
Plan to Share IPD: Undecided
HIPAA and CA regulations may prevent such sharing of data.